CLINICAL TRIAL: NCT03549832
Title: Sofosbuvir /Simeprevir/ Daclatasvir/Ribavirin Versus Sofosbuvir /Ombitasvir/ Paritaprevir /Ritonavir/Ribavirin in the Management of Hepatitis C Patients Fauilre to Prior Sofosbuvir/ Daclatasvir (An Open-labeled Randomized Trial)
Brief Title: Comparative Study of Two Regiemns in Management of Sofosbuvir/Daclatasvir Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Sohag University (Other); South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelsabour Mekky, Ass. Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17300204
Record Dates: First submitted 2018-05-27; First posted 2018-06-08 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: HCV Coinfection
Keywords: HCV; DAAs; Non-responder
MeSH Terms: interventions — Sofosbuvir; Simeprevir; daclatasvir; Ribavirin; ombitasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sof/sim/dac (Active Comparator): Sofosbuvir /Simeprevir/ Daclatasvir/Ribavirin
  Interventions: Drug: Sofosbuvir; Drug: Simeprevir; Drug: Daclatasvir; Drug: Ribavirin
- sof/omb/parit (Active Comparator): Sofosbuvir /Ombitasvir/ Paritaprevir /Ritonavir/Ribavirin
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin; Drug: Ombitasvir/paritaprevir/ritonavir

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg oral pills
Drug: Simeprevir — Simeprevir 150 mg oral pills
  Arms: sof/sim/dac
Drug: Daclatasvir — Daclatasvir 60 mg oral pills
  Arms: sof/sim/dac
Drug: Ribavirin — Ribavirin 200 mg oral pills
Drug: Ombitasvir/paritaprevir/ritonavir — Ombitasvir/paritaprevir/ritonavir oral pills
  Arms: sof/omb/parit

SUMMARY:
Now many cases reported failure to HCV treatment with Sofosbuvir/ Daclatasvir. retreat those patients is challenging. So, we aimed to Study the efficacy and safety of Sofosbuvir /Simeprevir/ Daclatasvir/Ribavirin versus Sofosbuvir /ombitasvir/ paritaprevir/ritonavir/ribavirin in the management of hepatitis C patients who failed to prior Sofosbuvir/ Daclatasvir regimens in an open-labeled randomized trial.

DETAILED DESCRIPTION:
HCV management with new DAAs is now promising. However, many cases reporting treatment failure either non-responder or relapse to HCV treatment with Sofosbuvir/ Daclatasvir. retreat those patients is challenging. So, we aimed to Study the efficacy and safety of Sofosbuvir /Simeprevir/ Daclatasvir/Ribavirin versus Sofosbuvir /ombitasvir/ paritaprevir/ritonavir/ribavirin in the management of hepatitis C patients who failed to prior Sofosbuvir/ Daclatasvir regimens in a multicenter open-labeled randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven CHC genotype 4
* 18 years old or more,
* prior HCV treatment failure to sofosbuvir /daclatasvir
* compensated liver disease.

Exclusion Criteria:

* Patients with combined HCV/HBV co-infection, hepatocellular carcinoma (HCC), decompensated liver cirrhosis (Child-Pugh score above 6), and non-genotype 4 were excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
SVR rate | 12 weeks
  The primary endpoint was the achievement of SVR at week 12 (SVR12) post-treatment. The potential adverse events were evaluated in each visit for the development of adverse events or any significant interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mekky, MD, Study Director — Assiut University
Locations (1):
- Assiut University Hopsital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gutierrez JA, Lawitz EJ, Poordad F. Interferon-free, direct-acting antiviral therapy for chronic hepatitis C. J Viral Hepat. 2015 Nov;22(11):861-70. doi: 10.1111/jvh.12422. Epub 2015 Jun 17. PMID 26083155